CLINICAL TRIAL: NCT00467051
Title: Treatment of Recurrent or Resistant Pediatric Malignant Germ Cell Tumors With Paclitaxel, Ifosfamide and Carboplatin
Brief Title: Combination Chemotherapy in Treating Young Patients With Recurrent or Resistant Malignant Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGCT0521; NCI-2009-00374 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AGCT0521; CDR0000542424; AGCT0521 (Other: Childrens Oncology Group); AGCT0521 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2015-03-20 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2017-10

CONDITIONS: Childhood Extracranial Germ Cell Tumor; Childhood Extragonadal Malignant Germ Cell Tumor; Childhood Malignant Ovarian Germ Cell Tumor; Childhood Malignant Testicular Germ Cell Tumor; Ovarian Choriocarcinoma; Ovarian Embryonal Carcinoma; Ovarian Yolk Sac Tumor; Recurrent Childhood Malignant Germ Cell Tumor; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Ovarian Germ Cell Tumor; Testicular Choriocarcinoma; Testicular Embryonal Carcinoma; Testicular Mixed Choriocarcinoma and Embryonal Carcinoma; Testicular Mixed Choriocarcinoma and Yolk Sac Tumor; Testicular Mixed Embryonal Carcinoma and Yolk Sac Tumor; Testicular Yolk Sac Tumor
MeSH Terms: conditions — Ovarian Germ Cell Cancer; Testicular Neoplasms; Carcinoma, Embryonal; Endodermal Sinus Tumor | interventions — Carboplatin; Filgrastim; Granulocyte Colony-Stimulating Factor; Ifosfamide; Paclitaxel; Taxes

ARMS (1):
- Treatment (chemotherapy, biological therapy) (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 1 hour on day 1 and ifosfamide IV over 1 hour on days 1-5. Beginning on day 6, patients receive filgrastim (G-CSF) subcutaneously or IV once daily until blood count returns to normal. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Biological: Filgrastim; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Biological: Filgrastim — Given IV or subcutaneously
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Other: Laboratory Biomarker Analysis — Optional correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This phase II trial is studying how well giving combination chemotherapy works in treating young patients with recurrent or resistant malignant germ cell tumors. Drugs used in chemotherapy, such as paclitaxel, ifosfamide, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate in pediatric patients with recurrent or resistant malignant germ cell tumors (GCT) treated with paclitaxel, ifosfamide, and carboplatin.

SECONDARY OBJECTIVES:

I. Determine the toxicity of this regimen in these patients. II. To Collect tissue for the tumor bank that will aid in the identification of the biological characteristics of recurrent GCT.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV over 3 hours and carboplatin IV over 1 hour on day 1 and ifosfamide IV over 1 hour on days 1-5. Beginning on day 6, patients receive filgrastim (G-CSF) subcutaneously or IV once daily until blood count returns to normal. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed (at original diagnosis) extracranial germ cell tumor (GCT) containing 1 of the following malignant elements:

  * Yolk sac tumor (endodermal sinus tumor)
  * Choriocarcinoma
  * Embryonal carcinoma
* Meets 1 of the following disease criteria:

  * Recurrent malignant disease
  * Chemotherapy-resistant disease
  * Relapsed disease
  * Disease refractory to conventional therapy
* Measurable disease
* Must have received a prior first-line chemotherapy regimen that included cisplatin
* Patients with tumor marker (AFP and/or BHCG) elevation alone or bone scan findings alone are not eligible*
* Patients with immature teratoma (any grade), germinoma, sex-cord stromal tumors, or recurrent GCT previously treated with surgery alone are not eligible
* Karnofsky performance status (PS) 50-100% (age > 16 years) OR Lansky PS 50-100% (age ≤ 16 years) OR ECOG PS 0-2
* Life expectancy ≥ 8 weeks
* Absolute neutrophil count ≥ 750/mm³
* Platelet count ≥ 75,000/mm³ (transfusion independent)
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR creatinine normal based on age/gender, as defined by the following:

  * ≤ 0.4 mg/dL (1 month to < 6 months of age)
  * ≤ 0.5 mg/dL (6 months to < 1 year of age)
  * ≤ 0.6 mg/dL (1 to < 2 years of age)
  * ≤ 0.8 mg/dL (2 to < 6 years of age)
  * ≤ 1.0 mg/dL (6 to < 10 years of age)
  * ≤ 1.2 mg/dL (10 to < 13 years of age)
  * ≤ 1.4 mg/dL (13 to ≥ 16 years of age) (female)
  * ≤ 1.5 mg/dL (13 to < 16 years of age) (male)
  * ≤ 1.7 mg/dL (≥ 16 years of age) (male)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) for age
* ALT < 2.5 times ULN for age
* Shortening fraction ≥ 27% by echocardiogram OR ejection fraction ≥ 50% by gated radionuclide study
* No dyspnea at rest
* No exercise intolerance
* Pulse oximetry > 94% (if there is clinical indication for determination)
* Patients with seizure disorder are eligible provided they are on non-enzyme inducing anticonvulsants and seizures are well controlled
* No CNS toxicity > grade 2
* No active graft-versus-host disease
* No allergy to Cremophor EL or castor oil
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent chemotherapy or immunomodulating agents
* Recovered from prior chemotherapy, immunotherapy, or radiotherapy
* At least 1 week since prior growth factors (2 weeks for pegfilgrastim)
* At least 1 week since prior biologic therapy
* At least 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosourea)
* At least 2 weeks since prior local palliative radiotherapy (i.e., small port)
* At least 6 months since prior craniospinal radiotherapy or radiotherapy to ≥ 50% of pelvis
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* At least 6 months since prior allogeneic stem cell transplantation
* Concurrent radiotherapy to localized painful lesions allowed provided at least 1 measurable lesion is not irradiated

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11-05 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Rodriguez-Galindo, Principal Investigator — Children's Oncology Group
Locations (95):
- United States (85):
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Harbor-University of California at Los Angeles Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health Richland, Columbia, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Carilion Clinic Children's Hospital, Roanoke, Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (8):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec
- San Jorge Children's Hospital, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Chemotherapy, Biological Therapy): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 1 hour on day 1 and ifosfamide IV over 1 hour on days 1-5. Beginning on day 6, patients receive filgrastim (G-CSF) subcutaneously or IV once daily until blood count returns to normal. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  paclitaxel: Given IV dosage 135 mg/m2/dose
  carboplatin: Given IV dosage in mg/m2 = Target AUC (mg•min/mL) x [(0.93 x GFR mL/min/m2) + 15]= 6.5 x [(0.93 x GFR mL/min/m2) + 15]. (BSA = body surface area in square meters). GFR is reported in institutions as "uncorrected" or "raw" (not normalized to BSA) or "corrected." This number needs to be converted to GFR in mL/min/m2.
  ifosfamide: Given IV dosage 1800 mg/m2/dose
  filgrastim: Given IV or subcutaneously dosage 1,080mg/m2/day divided to three equal doses of 360mg/m2
  laboratory biomarker analysis: Optional correlative studies
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Biological Therapy)
Started | 20
Completed | 18
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, Biological Therapy)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 13.5 [1 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 15
  Canada | 3
  Australia | 1
  Puerto Rico | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate as Measured by Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Patients who demonstrate a PR or CR, as defined below, will be considered as responders. RECIST criteria: CR (complete response) = disappearance of all target lesions, PR (partial response) = 30% decrease in the sum of the longest diameter of target lesions, PD (progressive disease) = 20% increase in the sum of the longest diameter of target lesions and SD (stable disease) = small changes that do not meet above criteria.
Time Frame: At baseline (day 1) and after completion of protocol therapy (2 cycles or 42 days)
Measure: Number; unit: participants
Arm/Group | Treatment (Chemotherapy, Biological Therapy)
Number analyzed (Participants) | 20
participants
  Responder | 12
  Non-Responder | 8

2. Secondary Outcome: The Number of Patients Who Experience at Least One Grade 3 or Higher CTC Version 4 Toxicity.
Time Frame: Two cycles of chemotherapy; expected to be 42 days of treatment.
Population: All eligible patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 20
Participants | 18

ADVERSE EVENTS:
Description: SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs.
Arm/Group | Treatment (Chemotherapy, Biological Therapy)
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 18/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Chemotherapy, Biological Therapy) (N=20)
Agitation (Psychiatric disorders) | 1
Alanine aminotransferase increased (Investigations) | 2
Anemia (Blood and lymphatic system disorders) | 8
Aspartate aminotransferase increased (Investigations) | 1
Ataxia (Nervous system disorders) | 1
Bladder infection (Infections and infestations) | 1
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1
Cardiac disorders - Other (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Infections and infestations - Other (Infections and infestations) | 4
Intracranial hemorrhage (Nervous system disorders) | 1
Lymphocyte count decreased (Investigations) | 5
Nail loss (Skin and subcutaneous tissue disorders) | 1
Nervous system disorders - Other (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 12
Oral hemorrhage (Gastrointestinal disorders) | 1
Platelet count decreased (Investigations) | 9
Vomiting (Gastrointestinal disorders) | 2
White blood cell decreased (Investigations) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.